CLINICAL TRIAL: NCT02556021
Title: A Multicenter, Double-blind, Randomized, Placebo-controlled Phase 3 Study to Evaluate the Efficacy and Safety of CJ-12420 in Patients With Non-erosive Reflux Disease
Brief Title: Study to Evaluate the Safety and Efficacy of CJ-12420 in Patients With Non Erosive Reflux Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: HK inno.N Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CJ_APA_302
Record Dates: First submitted 2015-09-16; First posted 2015-09-22 (Estimated); Last update posted 2018-04-04 (Actual); Status verified 2018-04

CONDITIONS: Non-erosive Reflux Disease
MeSH Terms: conditions — Non-Erosive Reflux Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- CJ-12420 50mg (Experimental): CJ-12420 50 mg, tablet, once daily, oral administration for up to 4 weeks
  Interventions: Drug: CJ-12420 50mg
- CJ-12420 100mg (Experimental): CJ-12420 100 mg, tablet, once daily, oral administration for up to 4 weeks
  Interventions: Drug: CJ-12420 100mg
- Placebo (Placebo Comparator): Placebo, tablet, once daily, oral administration for up to 4 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CJ-12420 50mg — CJ-12420 50mg, tablet, once daily, oral administration for up to 4 weeks
  Other Names: Not yet decided
  Arms: CJ-12420 50mg
Drug: CJ-12420 100mg — CJ-12420 100mg, tablet, once daily, oral administration for up to 4 weeks
  Other Names: Not yet decided
  Arms: CJ-12420 100mg
Drug: Placebo — Placebo, tablet, once daily, oral administration for up to 4 weeks
  Arms: Placebo

SUMMARY:
The purpose of this study is to demonstrate the superiority of efficacy of CJ-12420, once daily (QD), compared to placebo in patients with non-erosive reflux disease at Week 4

DETAILED DESCRIPTION:
This is a double blind, randomized, placebo-controlled, phase 3 study. Subjects will be randomly assigned to one of the three treatment groups (CJ-12420 50 mg or 100 mg or placebo).

All subjects will be asked to take two tablets at the same time each day throughout the study, and also all subjects will be asked to record daily symptom in a subject diary on a daily basis.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects aged between 20 and 75 years
2. Subjects who had experienced a minimum three-month history of main symptom(heartburn and regurgitation)
3. Subjects were to have normal esophagus confirmed by endoscopy within 14 days prior to randomization
4. Subjects who is able to understand and follow the instructions and is willing to participate throughout the entire study
5. Subjects who voluntarily signed written informed consent form
6. Subjects who agreed to use medically acceptable contraceptives during the period of study
7. Subjects who had experienced heartburn and regurgitation within 7 days before randomization. Entry into study also required that patients had experienced at least mild upper gastrointestinal symptoms on at least 2 days/week or at least moderate upper gastrointestinal symptoms on at least 1 day/week

Exclusion Criteria:

1. Subjects who cannot undergo EGD
2. Subjects who have esophageal stenosis, ulcer stenosis, gastroesophageal varices, Barrett's esophagus, active gastric ulcer, gastrointestinal bleeding or malignant tumor confirmed by EGD
3. Subjects who have erosive esophagitis, acute upper gastrointestinal bleeding, gastric ulcers or duodenal ulcers, acute erosive gastritis within 2 months before randomization. Subjects with gastric or duodenal erosions are allowed to be included.
4. Subjects who have warning symptoms of malignant gastrointestinal tract such as odynophagia, severe dysphagia, bleeding, weight loss, anemia, or bloody stool
5. Subjects with eosinophilic esophagitis
6. Subjects diagnosed with functional dyspepsia, primary esophageal motility disorder, IBS, IBD, etc. or with suspected IBS in the last 3 months
7. Subjects who have a history of gastric acid suppression surgery or upper gastrointestinal, esophageal surgery
8. Subjects who have bipolar disorder, anxiety disorder, panic disorder, somatoform disorder, personality disorder and psychiatric disorders.
9. Subjects who are taking antipsychotic drugs, antidepressants or antianxiety medications
10. Subjects who should continuously administer NSAIDs during the trial.
11. Pregnant or lactating women
12. Subjects with a history of clinically significant hepatic, renal, cardiovascular, respiratory, endocrine and CNS system disorder
13. Subjects with a history of hypersensitivity to the active ingredient or excipients of the study drug, etc.
14. Subjects who participated in the other clinical trial within 4 weeks prior to randomization

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 324 (Actual)
Dates: Start 2015-09-22; Primary Completion 2016-11-01 (Actual); Study Completion 2016-11-01 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with complete resolution of main symptoms (heartburn and regurgitation) at 4-week, defined as no episodes of symptom during the last 7 days of treatment, using Reflux Disease Questionnaire(RDQ) | 4 week

SECONDARY OUTCOMES:
Resolution of main symptoms(heartburn and regurgitation) at 2-week(for 7 consecutive days) | 2 week
RDQ score change | 4 week
Percentage of symptom free days | 4 week
  Symptom will be collected by patient diary.

CONTACTS AND LOCATIONS:
Locations (1):
- Yeouido St.Mary's Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kim SH, Cho KB, Chun HJ, Lee SW, Kwon JG, Lee DH, Kim SG, Jung HY, Kim JW, Lee JS, Park H, Choi SC, Jee SR, Kim HS, Ko KH, Park SJ, Lee YC, Park SH, Kim AR, Kim EJ, Park HW, Kim BT, Song GS. Randomised clinical trial: comparison of tegoprazan and placebo in non-erosive reflux disease. Aliment Pharmacol Ther. 2021 Aug;54(4):402-411. doi: 10.1111/apt.16477. Epub 2021 Jul 6. PMID 34227708